CLINICAL TRIAL: NCT01157936
Title: Effect of Hyperuricemia Treatment on Hypertension and Metabolic Syndrome
Brief Title: Hyperuricemia on Hypertension and Metabolic Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Instituto Nacional de Cardiologia Ignacio Chavez (Other)
Collaborators: National Council of Science and Technology, Mexico (Other)
Responsible Party: Principal Investigator, Magdalena Madero, Chief Nephrology Division, Instituto Nacional de Cardiologia Ignacio Chavez
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: HYPERURICEMIA 2010; ALOPURINOL (Other: ALUPORINOL)
Record Dates: First submitted 2010-07-07; First posted 2010-07-08 (Estimated); Last update posted 2014-07-24 (Estimated); Status verified 2014-07

CONDITIONS: Systolic and Diastolic Blood Pressure Levels; Uric Acid Levels; Metabolic Syndrome Parameters; Hepatic Enzymes
Keywords: hypertension; hyperuricemia; metabolic syndrome
MeSH Terms: conditions — Systolic Murmurs; Hypertension; Hyperuricemia; Metabolic Syndrome | interventions — Allopurinol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Allopurinol treatment (Active Comparator)
  Interventions: Drug: Allopurinol
- Placebo (Placebo Comparator)
  Interventions: Other: placebo

INTERVENTIONS:
Drug: Allopurinol — daily dosage
  Other Names: xanthine oxidase inhibitor
  Arms: Allopurinol treatment
Other: placebo — daily dosage
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the influence of hyperuricemia treatment compared with placebo on participants with high risk of hypertension and metabolic syndrome.

DETAILED DESCRIPTION:
Elevated consumption of high fructose corn syrup has lead to an increase of 30% of fructose intake since the last 20 years. Important data supporting this fact can be reflected on incidence and prevalence of Metabolic syndrome and hyperuricemia.

A peculiar effect of fructose intake demonstrated in animal models is the development of elevated uric acid levels; also some studies have found a clear association between hyperuricemia as an important risk factor for hypertension, diabetes mellitus, chronic kidney disease and metabolic syndrome.

Taking into account the existing evidence, our clinical research team presents this protocol as a way to evaluate the effect of uric acid treatment and its relation with Fructose consumption, metabolic syndrome parameters, hyperuricemia and risk of hypertension.

Confirming evidence with clinical basis may be the initial strategy to create primary prevention programs to control this health problems affecting Mexican Population.

ELIGIBILITY:
Inclusion Criteria:

* adults with blood pressure from 120/80 mmHg and less than 140/90 mmHg
* no pharmacological treatment for blood pressure control

Exclusion Criteria:

* hypertension (more than 140/90mmHg)
* Diabetes Mellitus type 1 or 2
* Chronic kidney disease (MDRD less than 60)
* Hepatic Disease
* Malignancy
* Pregnancy
* patient receiving any medication

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2010-07; Primary Completion 2011-02 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Effect of hyperuricemia treatment on systemic blood pressure | 14 weeks
  participants will be randomized to a 4 week placebo versus alopurinol treatment followed by a wash out period. After crossover them, they will receive the complementary pharmacological intervention for another 4 weeks.

SECONDARY OUTCOMES:
Effect of hyperuricemia treatment on metabolic syndrome parameters | 14 weeks
  baseline and final laboratory samples during pre and post crossover periods will include metabolic syndrome measurements (triglycerides, cholesterol, glucose and abdominal perimeter).

CONTACTS AND LOCATIONS:
Overall Officials: Magdalena Madero, MD, Principal Investigator — Instituto Nacional de Cardiología Ignacio Chávez
Locations (1):
- Insituto Nacional de Cardiología Ignacio Chávez, México, State of Mexico, Mexico

REFERENCES:
- [Derived] Fravel MA, Ernst ME. Management of gout in the older adult. Am J Geriatr Pharmacother. 2011 Oct;9(5):271-85. doi: 10.1016/j.amjopharm.2011.07.004. Epub 2011 Aug 17. PMID 21849262